CLINICAL TRIAL: NCT07081919
Title: Effectiveness, Stability and Influence Factors of Femtosecond Laser Assisted Cataract Surgery
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jin Yang, Chief Physician, Eye & ENT Hospital of Fudan University
Other Study IDs: FSAK during cataract surgery
Record Dates: First submitted 2025-06-01; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Corneal Astigmatism; Cataract
Keywords: femtosecond laser-assisted arcuate keratotomy; cataract surgery; corneal astigmtism; astigmatism treatment stability; predictors of surgical outcomes
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FSAK with Cataract Surgery: Participants in this group undergo femtosecond laser-assisted arcuate keratotomy (FSAK) combined with standard cataract surgery
  Interventions: Procedure: femtosecond laser-assisted arcuate keratotomy (FSAK) combined with standard cataract surgery

INTERVENTIONS:
Procedure: femtosecond laser-assisted arcuate keratotomy (FSAK) combined with standard cataract surgery — 1. 5-year follow-up assessing stability of astigmatism correction. Most FSAK studies track ≤2 years. This addresses critical evidence gaps in durability
  2. Combines topographic data with patient-reported visual function (VF-14/QoV questionnaires at all visits. Links anatomical changes to real-world visual experiences

SUMMARY:
What is this study about? This study looks at whether a laser procedure called femtosecond laser-assisted arcuate keratotomy (FSAK) helps people with both cataracts and mild astigmatism see more clearly after cataract surgery. Astigmatism causes blurry vision because the front of the eye (cornea) is curved unevenly. The FSAK procedure uses a computer-guided laser to make tiny, precise cuts in the cornea during cataract surgery to fix this curve. the investigators want to see if this improves vision long-term (up to 5 years) and what factors affect how the investigatorsll it works.

Who can join? the investigators are looking for adults aged 20-80 years who:

Have cataracts and mild-to-moderate astigmatism (0.75-2.0 diopters) Plan to have cataract surgery Have not had prior eye surgeries (like LASIK) Do not have severe dry eye or other eye diseases (like glaucoma or retina problems) What will happen in the study?

Surgery: Participants will have cataract surgery combined with the FSAK procedure. The surgeon uses a laser to make tiny curved cuts in the cornea to reshape it.

Follow-up visits: Participants will have regular eye check-ups for 5 years after surgery. These include:

Vision tests (reading eye charts) Measurements of the eye's shape using painless imaging machines Questionnaires about vision quality and daily activities Time commitment: Visits happen at 1 the investigatorsek, 1 month, 3 months, 6 months, 1 year, 2 years, and 5 years after surgery. Each visit takes about 1-2 hours.

Why is this study important? FSAK may help people with astigmatism see clearly after cataract surgery without needing glasses as often. By tracking results for 5 years, the investigators'll learn how long the benefits last and who benefits most. This could help doctors better personalize treatment in the future.

Who is running the study? Eye doctors at Fudan University Eye & ENT Hospital (Shanghai) and Shanghai Peace Eye Hospital. About 105 people will take part.

DETAILED DESCRIPTION:
Study Description for General Audience

What's the problem? Many people with cataracts also have an irregularly curved front surface of the eye (called astigmatism). After cataract surgery, this astigmatism can still cause blurry or distorted vision, making everyday tasks like reading or driving difficult. While glasses or special lenses can help, many hope to reduce their dependence on them after surgery.

What's being tested?

This study evaluates a laser procedure called Femtosecond Laser-Assisted Arcuate Keratotomy (FSAK). During cataract surgery:

A computer-guided laser makes tiny, curved incisions in the cornea (the eye's clear front window).

These precise incisions gently reshape the cornea to improve its natural curve. Think of it like a sculptor smoothing uneven surfaces-but using light-speed technology.

Why is this study unique?

While FSAK isn't brand new, the investigators lack long-term data on:

How the investigatorsll it holds up over 5+ years. Which factors predict success (e.g., does participantsr eye's shape or pressure affect results?).

the investigators're following participants for 5 years to ansthe investigatorsr these questions-far longer than most existing studies.

What will participants experience?

Surgery: FSAK is combined with standard cataract removal. The laser step adds only minutes.

Follow-ups: Painless check-ups at 1 the investigatorsek, 1 month, 3 months, 6 months, 1 year, 2 years, and 5 years after surgery. These involve:

Reading eye charts. Quick scans to map the eye's surface. Short questionnaires about vision quality (e.g., glare at night or reading small print).

Why does this matter?

If successful, FSAK could:

* Help people see clearly longer after cataract surgery.
* Reduce the need for glasses or contacts.
* Give doctors better tools to personalize treatment.

Who's involved?

Led by eye specialists at Fudan University Eye & ENT Hospital and Shanghai Peace Eye Hospital.

ELIGIBILITY:
Inclusion Criteria

* Age: 20-80 years
* Age-related cataracts
* Regular corneal astigmatism (0.75-2.0 diopters) confirmed by Pentacam/IOLMaster 700
* Surgical Plan: Scheduled for femtosecond laser-assisted cataract surgery
* Central corneal thickness ≥500 µm
* Endothelial cell count ≥2,000 cells/mm²
* Best-corrected visual acuity (BCVA) improvable to ≥20/40

Exclusion Criteria

* Prior corneal refractive surgery (e.g., LASIK, PRK)
* Intraocular surgery (e.g., glaucoma filtering surgery)
* Irregular astigmatism (keratoconus, scarring, post-traumatic distortion)
* Active ocular inflammation or infection
* Corneal endothelial disease (e.g., Fuchs' dystrophy)
* Severe dry eye (Schirmer test ≤5 mm/5 min)
* Uncontrolled glaucoma (IOP >21 mmHg on medication)
* Macular pathology (e.g., AMD, DME affecting visual potential)
* Amblyopia
* Autoimmune diseases affecting cornea (e.g., rheumatoid arthritis, Sjögren syndrome)
* Diabetes mellitus with retinopathy
* Pregnancy/Lactation
* Inability to complete 5-year follow-up

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with regular corneal astigmatism of 0.75-2.0 D who plan to undergo cataract surgery.
  Aged between 20 and 80 years old.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2030-04-22 (Estimated); Study Completion 2031-04-22 (Estimated)

PRIMARY OUTCOMES:
Change in corneal astigmatism magnitude (diopters) from baseline | Preoperative; 1 week postoperatively, 1 month postoperatively, 3 months postoperatively, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively

SECONDARY OUTCOMES:
Visual Acuity-UCVA | Preoperative; 1 week postoperatively, 1 month postoperatively, 3 months postoperatively, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively
  Uncorrected Distance Visual Acuity (UDVA) at 5m (logMAR)
Visual acuity-BCVA | Preoperative; 1 week postoperatively, 1 month postoperatively, 3 months postoperatively, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively
  Best-Corrected Visual Acuity (BCVA) at 5m (logMAR)
Manifest refraction spherical equivalent (MRSE) in Diopter (D) | Preoperative; 1 week postoperatively, 1 month postoperatively, 3 months postoperatively, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively
Corneal Topography | Preoperative; 1 week postoperatively, 1 month postoperatively, 3 months postoperatively, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively
  Corneal Topography assesses corneal curvature, with data collected using the Pentacam instrument and IOL Master. The measured outcome reflects the corneal's refractive power and shape characteristics. Corneal curvature is reported in diopters (D) , a standard unit for quantifying refractive power in ophthalmic measurements.
Objective Optical Quality | Preoperative; 1 week postoperatively, 1 month postoperatively, 3 months postoperatively, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively
  Objective visual quality is evaluated by measuring Total ocular higher - order aberrations (HOAs, unit: µm) and Strehl ratio (SR) using the iTrace instrument. Total ocular higher - order aberrations reflect the deviation of the eye's optical system from an ideal state, where higher values generally indicate greater optical imperfections that may disrupt visual clarity. The Strehl ratio, on the other hand, quantifies the quality of optical imaging; a higher SR (ranging from 0 to 1, with 1 representing ideal optical quality) signifies better visual quality, as it relates to the concentration of light in the retinal image. These metrics, derived from iTrace measurements, provide objective assessments of how well the eye processes visual input, crucial for evaluating surgical outcomes (e.g., cataract or refractive surgery) and ocular health.
Patient-Reported Outcomes | Preoperative; 1 week postoperatively, 1 month postoperatively, 3 months postoperatively, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively
  bjective visual quality can be assessed with the Visual Function-14 (VF-14) questionnaire, which evaluates 14 vision-dependent daily activities. Patients self-rate their functional limitations, with scores ranging from 0 (worst) to 100 (best), where higher scores indicate better visual function. It is administered preoperatively and 3 months postoperatively to measure changes, with a minimal clinically important difference of 15.57, meaning a score change exceeding this value signifies a meaningful improvement The DOI of reference for visual function questionnaire is 10.1016/j.ophtha.2010.04.009.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye and Ear, Nose, and Throat Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data contain sensitive biometric identifiers (e.g., corneal topography maps) that cannot be fully de-identified